CLINICAL TRIAL: NCT03237143
Title: Quality of Erections After Completing a Low-intensity Extracorporeal Shock Wave Treatment Cycle
Brief Title: Low-intensity Extracorporeal Shock Wave for Erectile Disfunction
Status: Terminated | Type: Observational
Why Stopped: The research question was resolved in a metanalysis
Sponsor: Boston Medical Group (Industry)
Responsible Party: Sponsor
Other Study IDs: BMGC-1
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2017-08

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Erectile dysfunction occurs in a high percentage of patients today, showing not only an association with various pathologies but also frequent refractoriness to conventional pharmacological treatment options such as monotherapy. The objective of this study is to evaluate the response to low-intensity extracorporeal shock wave therapy in a group of patients with organic vascular erectile dysfunction with a history of more than three months.

Materials and Methods: Observational retrospective study. The researchers reviewed clinical records of patients with a clinical diagnosis of organic vascular erectile dysfunction (ED) of more than 3 months duration, who received 5 outpatient shock wave therapy sessions, in the male sexual health clinics of the Boston Medical Group from Spain and Mexico. The patients were evaluated with the erection hardness score (EHS) before the first session, at the end of the last session and one month after the last session.

DETAILED DESCRIPTION:
Clinical records of patients over 18 years of age with a clinical diagnosis of organic vascular ED, of more than three months and with an erection hardness score (EHS)(17) of three or less, treated between April 2014 and February 2015 in the Boston Medical Group male sexual health clinics of twelve cities in Spain (Madrid, Barcelona, Valencia, Seville, Coruña, Bilbao, Malaga, Zaragoza, Murcia, Alicante, Cordoba and Jerez) and four in Mexico (Altavista, Reforma, Monterrey and Naucalpan), were reviewed. The researchers excluded patients with ED caused by side effects from drugs or spinal cord injury; situational ED (obvious psychological origin); lesions, loss of skin or penile implant; and patients who did not adequately complete the LI-ESWT (Low-intensity extracorporeal shock wave therapy).

After the initial assessment and diagnosis consultation, each patient received a treatment of 5 sessions (1 session per week) of 20 minutes of LI-ESWT, carried out with the DUOLITH SD1 (Storz Tägerwilen, Switzerland). They received 3,000 impulses per session at 0.1 mJ/mm2, divided over six sites, four on the penis and two on the crura. All sessions were outpatient visits and no anaesthetic was used. The EHS for all patients was measured at three stages: before the first session, at the end of the last session (5 weeks after the first session) and one month after the last session. When patients were receiving concomitant drug treatment for their dysfunction, they were asked to indicate their perception free of the effect thereof. All the clinical information was recorded by qualified physicians on a standardised form using centralised software on a secure server.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* clinical diagnosis of organic vascular ED of more than three months and with an erection hardness score (EHS) of three or less

Exclusion Criteria:

* patients with ED caused by side effects from drugs or spinal cord injury
* situational ED (obvious psychological origin)
* lesions, loss of skin or penile implant
* patients who did not adequately complete the LI-ESWT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated between April 2014 and February 2015 in the Boston Medical Group male sexual health clinics of twelve cities in Spain (Madrid, Barcelona, Valencia, Seville, Coruña, Bilbao, Malaga, Zaragoza, Murcia, Alicante, Cordoba and Jerez) and four in Mexico (Altavista, Reforma, Monterrey and Naucalpan)
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Erection hardness score | one month after the last session
  Erection hardness score (EHS)

SECONDARY OUTCOMES:
Erection hardness score | At the end after the last session
  Erection hardness score (EHS)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayala HAC, Cuartas JPS, Cleves DC. Impact on the Quality of Erections after Completing a Low-Intensity Extracorporeal Shock Wave Treatment Cycle on a Group of 710 Patients. Adv Urol. 2017;2017:1843687. doi: 10.1155/2017/1843687. Epub 2017 Dec 21. PMID 29430250